CLINICAL TRIAL: NCT05563012
Title: Single-arm Phase II Clinical Study of Short-course Radiotherapy Combined With Neoadjuvant Chemotherapy and PD-1 Inhibitor in the Treatment of Locally Advanced Gastric Adenocarcinoma
Brief Title: Short-course Radiotherapy Combined With Neoadjuvant Chemotherapy and PD-1 Inhibitor in the Treatment of Locally Advanced Gastric Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Xiangpan Li, Professor, Renmin Hospital of Wuhan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WDRY2022-KI78
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Disorder in Complete Remission in Response to Treatment
MeSH Terms: interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with untreated, operable locally advanced gastric adenocarcinoma (Experimental): Drug: Sintilimal Injection Sintilimal (200mg) will be given i.v. on day 1 of each 3-week cycle.
  Drug: Capecitabine Capecitabine (1000mg/m2) will be administered orally twice daily on days 1-14 of each 3-week cycle.
  Drug: Oxaliplatin Oxaliplatin (130mg/m2) will be given i.v. on day 1 of each 3-week cycle.
  Interventions: Drug: Sintilimal Injection

INTERVENTIONS:
Drug: Sintilimal Injection — Sintilimal (200mg) will be given i.v. on day 1 of each 3-week cycle.
  Other Names: Capecitabine; Oxaliplatin

SUMMARY:
This is a Prospective, Single-center, Single-arm, phase II clinical trial to explore the efficacy and safety of sintilimab (PD1 inhibitor) combined with XELOX chemotherapy, evaluate the pathological complete response rate of short-course radiotherapy combined with sintilimab and XELOX chemotherapy in neoadjuvant therapy for locally advanced gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. All individuals recruited signed a written informed consent;
2. Aged between 18 and 75 years;
3. Histologically confirmed gastric adenocarcinoma, and Stage III (cT3-4aN1-3 M0, American Joint Committee on Cancer (AJCC) TNM staging system 8th edition) gastric cawas confirmed by enhanced CT/MRI scan (endoscopic ultrasonography (EUS) and laparoscopic exploration if necessary), and the lesion was resectable;
4. No previous systemic therapy, including including surgery, radiotherapy, chemotherapy and immunotherapy, etc；
5. Patients who have no contraindications and consent to radical surgery;
6. Eastern Cooperative Group (ECOG) performance status score 0 or 1;
7. Expected survival time > 6 months;
8. The main organ function of cases should be normal, and meet the following criteria: ①Absolute neutrophil count (ANC)≥1.5×109/L (no Granulocyte colony-stimulating factor within 14 days prior to enrolment); ②Platelets ≥100×109/L (no blood transfusion within 14 days prior to enrolment); ③Hemoglobin>90g/L (no blood transfusion or no erythropoietin (EPO) dependence within 14 days prior to enrolment); ④Total bilirubin (TBIL) ≤1.5 x upper limit of normal (ULN), such as total bilirubin > 1.5 x ULN but direct bilirubin ≤1.5 x ULN was also allowed to be enrolled; ⑤ALT (glutamic-pyruvic transaminase) and AST (glutamic-oxalacetic transaminase) ≤2.5 × ULN; ⑥Serum Cr≤1.5 × ULN and creatinine clearance ≥60 ml/min (Cockcroft-Gault formula); ⑦International normalized ratio (INR) <1.5 or prothrombin time (PT)≤1.5 ULN; ⑧Thyroid stimulating hormone (TSH) was normal. If TSH was abnormal, subjects with total T3 (or FT3) and FT4 normal could also be enrolled; ⑨Myocardial infarction was normal.
9. Female subjects of reproductive age must conduct pregnancy test (serum or urine) within 3 days before the first study drug administration (day 1 of cycle 1), and the results are negative. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as those who had been postmenopausal for at least 1 year or who had undergone surgical sterilization or hysterectomy;
10. If there was a risk of conception, all subjects (male or female) were required to use contraception with an annual failure rate of less than 1% for the entire treatment period until 120 days after the last administration of the test drugs (or 180 days after the last administration of the chemotherapy drug ).

Exclusion Criteria:

1. Other malignancy disease history within five years, with the exception of basal cell carcinoma or squamous carcinoma of skin, and carcinoma in situ that have undergone radical resection;
2. Endoscopic signs of active bleeding in the lesion;
3. Is participating in an interventional clinical study or has received another study drug or used a study device within 4 weeks before the first study drug administration;
4. Prior treatment with an anti-PD-1, anti-PD-L1 or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g. CTLA-4, OX40, CD137) drugs;
5. Systemic systemic therapy with Chinese patent drugs or immunomodulatory agents (including thymosin, interferon, and interleukin, except for local use to control pleural effusion) with anti-tumor indications was received within 2 weeks before the first study drug administration;
6. Active autoimmune disease requiring systemic therapy (e.g., use of disease-modifying agents, glucocorticoids, or immunosuppressants) occurred within 2 years before the first study drug administration. Replacement therapy (e.g., thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) is not considered a form of systemic treatment;
7. Had received systemic glucocorticoid therapy (excluding nasal, inhaled, or other local glucocorticoids) or any other form of immunosuppressive therapy within 7 days before the first study drug administration;
8. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
9. Known allergy to drugs used in this study;
10. Unable to intake Capecitabine orally (such as the inability to swallow and intestinal obstruction);
11. Failure to recover from treatment-related toxicity/complications to baseline or grade-1 AEs (except for fatigue and hair loss);
12. Has a known history of HIV infection (HIV 1/2 antibody positive);
13. Untreated active hepatitis B (defined as HBsAg-positive with a detected HBV-DNA copy number greater than the upper limit of normal values in the laboratory at the study center); Note: Hepatitis B subjects who meet the following criteria can also be enrolled: ①With HBV viral load <1000 copies /ml (200 IU/ml) before the first study drug administration, subjects should receive anti-HBV therapy to avoid virus reactivation throughout the study chemotherapy drug treatment; ②For subjects with anti-HBC (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but monitoring of viral reactivation is required;
14. Active HCV-infected subjects (HCV antibody positive with HCV-RNA levels higher then the lower limit of detection);
15. Had received live vaccine within 30 days before the first study drug administration; Note: Inactivated virus vaccine for injection against seasonal influenza is permitted for 30 days before the first study drug administration; However, live attenuated influenza vaccines administered intranasally are not allowed;
16. Pregnant or lactating women;
17. The presence of any severe or uncontrolled systemic disease, e.g; ①The resting ECG showed significant abnormalities in rhythm, conduction or morphology with severe symptoms and difficult to control, such as complete left bundle branch block, degree ⅱ higher heart block, ventricular arrhythmia or atrial fibrillation; ②Unstable angina pectoris, congestive heart failure, New York Heart Association (NYHA) grade ≥ 2 chronic heart failure; ③Any arterial thrombosis, embolism, or ischemia, such as myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, occurred in the 6 months prior to enrollment; ④Poor blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg); ⑤Has a history of noninfectious pneumonia requiring glucocorticoid therapy within 1 year before the first study drug administration or active interstitial lung disease; ⑥Active pulmonary tuberculosis; ⑦Have active or uncontrolled infections requiring systemic therapy; ⑧There are active diverticulitis, abdominal abscess, and gastrointestinal obstruction; ⑨Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; ⑩Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L); ⑪Urine routine indicated urinary protein ≥++, and 24-hour urinary protein > 1.0 g on urine dipstick; ⑫Patients with mental disorders who are unable to actively cooperate with treatment;
18. Subjects are not eligible to participate in the study if they have abnormal medical history or evidence of disease, treatment or laboratory test values that may interfere with the results of the trial or prevent their full participation in the study, or if they have other conditions or potential risks that the investigator considers inappropriate for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | 36 months
  Defined as lack of any viable tumor cells in the surgically removed tumor and lymph node tissues.

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | 36 months
  Defined as the proportion of subjects with 10% or less of residual viable tumor cells in the resected primary tumor.
Disease-free survival (DFS) | 36 months
  Defined as the time from surgery to the time of first recurrence or death, whichever occurred first.
overall survival (OS) | 36 months
  OS is the time from enrollment to death due to any cause. OS is the time from enrollment to death due to any cause. OS is the time from enrollment to death due to any cause.OS is the time from enrollment to death due to any cause.
  OS is the time from enrollment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangpan Li, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China